CLINICAL TRIAL: NCT03951753
Title: The Effect of Tirzepatide on α and β Cell Function and Insulin Sensitivity in Patients With Type 2 Diabetes Mellitus
Brief Title: A Study of Tirzepatide in Participants With Type 2 Diabetes Mellitus (T2DM)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: 17091; I8F-MC-GPGT (Other: Eli Lilly and Company); 2018-003343-37 (EudraCT Number)
Record Dates: First submitted 2019-05-14; First posted 2019-05-15 (Actual); Results first posted 2023-03-20 (Actual); Last update posted 2023-03-20 (Actual); Status verified 2022-06

CONDITIONS: Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Tirzepatide; semaglutide

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (3):
- Tirzepatide 15 mg (Experimental): Participants received 15 milligram (mg) tirzepatide administered subcutaneously (SC) once weekly for 28 weeks.
  Interventions: Drug: Tirzepatide
- Semaglutide 1 mg (Active Comparator): Participants received 1 mg Semaglutide administered SC once weekly for 28 weeks.
  Interventions: Drug: Semaglutide
- Placebo (Placebo Comparator): Participants received Placebo administered SC once weekly for 28 weeks.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Tirzepatide — Administered SC
  Other Names: LY3298176
  Arms: Tirzepatide 15 mg
Drug: Semaglutide — Administered SC
  Arms: Semaglutide 1 mg
Drug: Placebo — Administered SC
  Arms: Placebo

SUMMARY:
This is a study for participants with type 2 diabetes mellitus. The main purpose of this study is to learn more about how tirzepatide, semaglutide and placebo affect the body's ability to respond to blood sugar levels after a meal. The study will last up to 40 weeks, including a 28-week treatment period.

ELIGIBILITY:
Inclusion Criteria:

* Have T2DM for at least 6 months
* Treated with diet and exercise and stable dose(s) of metformin, with or without 1 additional stable dose of oral antihyperglycemia medication other than metformin, 3 months prior to study entry
* Have a hemoglobin A1c (HbA1c) value at screening of ≥7% and ≤ 9.5 % if on metformin only; or ≥6.5% and ≤9.0% if on metformin in combination with oral antihyperglycemia medications other than metformin
* Have a body mass index (BMI) between 25 and 45 kilograms per square meter (kg/m² ) inclusive, at screening; are of stable weight (±5%) >3 months prior to screening

Exclusion Criteria:

* Have a history of proliferative retinopathy or maculopathy as determined by the investigator based on a recent (<1.5 years) ophthalmologic examination
* Impaired renal estimated glomerular filtration rate (eGFR) <45 milliliters per minute per 1.73 square meters (mL/min/1.73 m²) calculated by Chronic Kidney Disease Epidemiology Collaboration (CKD-EPI)
* Have a history or current cardiovascular, respiratory, hepatic, renal, GI,endocrine, hematological or neurological disorders capable of significantly altering the absorption, metabolism or elimination of drugs; of constituting a risk when taking the study drug; or of interfering with the interpretation of data

Ages: 20 Years to 74 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 117 (Actual)
Dates: Start 2019-06-28 (Actual); Primary Completion 2021-04-08 (Actual); Study Completion 2021-04-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (2):
- Germany (2):
  - Profil Institut für Stoffwechselforschung, Neuss, North Rhine-Westphalia
  - Profil Mainz GmbH & Co. KG, Mainz, Rhineland-Palatinate

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Heise T, DeVries JH, Urva S, Li J, Pratt EJ, Thomas MK, Mather KJ, Karanikas CA, Dunn J, Haupt A, Milicevic Z, Coskun T. Tirzepatide Reduces Appetite, Energy Intake, and Fat Mass in People With Type 2 Diabetes. Diabetes Care. 2023 May 1;46(5):998-1004. doi: 10.2337/dc22-1710. PMID 36857477
- [Derived] Heise T, Mari A, DeVries JH, Urva S, Li J, Pratt EJ, Coskun T, Thomas MK, Mather KJ, Haupt A, Milicevic Z. Effects of subcutaneous tirzepatide versus placebo or semaglutide on pancreatic islet function and insulin sensitivity in adults with type 2 diabetes: a multicentre, randomised, double-blind, parallel-arm, phase 1 clinical trial. Lancet Diabetes Endocrinol. 2022 Jun;10(6):418-429. doi: 10.1016/S2213-8587(22)00085-7. Epub 2022 Apr 22. PMID 35468322

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Tirzepatide 15 mg | Semaglutide 1 mg | Placebo
Started | 45 | 44 | 28
Completed | 41 | 43 | 24
Not Completed | 4 | 1 | 4
Not completed — Adverse Event | 1 | 0 | 3
Not completed — Withdrawal by Subject | 3 | 1 | 0
Not completed — Lost to Follow-up | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Population: All randomized participants who received at least one dose of study drug.
Groups:
- Tirzepatide 15 mg: Participants received 15 mg Tirzepatide administered SC once weekly for 28 weeks.
- Total: Total of all reporting groups
Arm/Group | Tirzepatide 15 mg | Semaglutide 1 mg | Placebo | Total
Number analyzed (Participants) | 45 | 44 | 28 | 117
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 31 | 20 | 18 | 69
  >=65 years | 14 | 24 | 10 | 48
Age, Continuous [Mean (Standard Deviation); unit: years] | 61.1 (7.1) | 63.7 (5.9) | 60.4 (7.6) | 61.9 (6.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14 | 10 | 7 | 31
  Male | 31 | 34 | 21 | 86
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 45 | 44 | 28 | 117
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 1 | 0 | 0 | 1
  White | 44 | 44 | 28 | 116
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  Germany | 45 | 44 | 28 | 117
HbA1c (%) [Mean (Standard Deviation); unit: percentage] — HbA1c is the glycosylated fraction of hemoglobin A. HbA1c is measured primarily to identify average plasma glucose concentration over prolonged periods of time.
  percentage | 7.83 (0.72) | 7.70 (0.60) | 7.90 (0.51) | 7.80 (0.63)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Total Clamp Disposition Index (cDI)
Description: cDI is defined as the product of the M-value derived from the hyperinsulinemic euglycemic clamp over the last 30 minutes and total insulin secretion (ISR AUC0-120min) derived from the insulin secretion rate based on C-peptide using the using the deconvolution technique divided by the total glucose AUC0-120min from the hyperglycemic clamp portion of the study. Least squares (LS) mean was determined by analysis of covariance (ANCOVA) model for endpoint measures: log(Actual Measurement/Baseline) = log(Baseline) + Treatment (Type III sum of squares).
Time Frame: Baseline, Week 28
Population: All randomly assigned participants who received at least 1 dose of study drug and have evaluable data.
Measure: Least Squares Mean (Standard Error); unit: pmol*m-2*L*min-2*kg-1
Arm/Group | Tirzepatide 15 mg | Semaglutide 1 mg | Placebo
Number analyzed (Participants) | 39 | 39 | 24
pmol*m-2*L*min-2*kg-1 | 1.9 (0.16) | 1.1 (0.10) | 0.0 (0.03)
Statistical Analysis 1: Comparison: Semaglutide 1 mg vs Placebo; Test type: Other; p < 0.001, ANCOVA; Data were analysed with ANCOVA in log transformed data; Least Squares Mean Difference = 1.08, 95% CI 2-sided [0.87 to 1.29], Standard Error of Mean 0.107 — Data were analysed with ANCOVA in log transformed data. Results were converted back to original scale
Statistical Analysis 2: Comparison: Tirzepatide 15 mg vs Placebo; Test type: Other; p < 0.001, ANCOVA; Data were analysed with ANCOVA in log transformed data; Least Squares Mean Difference = 1.92, 95% CI 2-sided [1.59 to 2.24], Standard Error of Mean 0.166 — Data were analysed with ANCOVA in log transformed data. Results were converted back to original scale
Statistical Analysis 3: Comparison: Tirzepatide 15 mg vs Semaglutide 1 mg; Test type: Other; p < 0.001, ANCOVA; Data were analysed with ANCOVA in log transformed data; Least Squares Mean Difference = 0.84, 95% CI 2-sided [0.46 to 1.21], Standard Error of Mean 0.192 — Data were analysed with ANCOVA in log transformed data. Results were converted back to original scale

2. Secondary Outcome: Change From Baseline in Fasting Glucose
Description: Fasting glucose is a test to determine sugar levels in blood sample after an overnight fast. Fasting glucose was measured prior to standardized mixed-meal tolerance tests (sMMTT). LS mean was determined by ANCOVA model for endpoint measures: Variable = Baseline + Treatment (Type III sum of squares).
Time Frame: Baseline, Week 28
Population: All randomly assigned participants who received at least 1 dose of study drug and have evaluable data.
Measure: Least Squares Mean (Standard Error); unit: milligrams per decilitre (mg/dL)
Arm/Group | Tirzepatide 15 mg | Semaglutide 1 mg | Placebo
Number analyzed (Participants) | 41 | 43 | 24
milligrams per decilitre (mg/dL) | -51.4 (2.30) | -42.4 (2.22) | -4.3 (2.98)
Statistical Analysis 1: Comparison: Semaglutide 1 mg vs Placebo; Test type: Other; p < 0.001, ANCOVA; Least Squares Mean Difference = -38.1, 95% CI 2-sided [-45.4 to -30.7]
Statistical Analysis 2: Comparison: Tirzepatide 15 mg vs Placebo; Test type: Other; p < 0.001, ANCOVA; Least Squares Mean Difference = -47.1, 95% CI 2-sided [-54.6 to -39.5]
Statistical Analysis 3: Comparison: Tirzepatide 15 mg vs Semaglutide 1 mg; Test type: Other; p = 0.006, ANCOVA; Least Squares Mean Difference = -9.0, 95% CI 2-sided [-15.4 to -2.6]

3. Secondary Outcome: Change From Baseline in Postmeal Glucose
Description: Total AUC from time zero to 240 minutes after start of the meal [AUC0-240min]) during sMMTT was evaluated. LS mean was determined by ANCOVA model for endpoint measures: Variable = Baseline + Treatment (Type III sum of squares) and ANOVA model for baseline measures: Variable = Treatment (Type III sum of squares).
Time Frame: Baseline, Week 28
Population: All randomly assigned participants who received at least 1 dose of study drug and have evaluable data.
Measure: Least Squares Mean (Standard Error); unit: Milligrams per decilitre*minute
Arm/Group | Tirzepatide 15 mg | Semaglutide 1 mg | Placebo
Number analyzed (Participants) | 41 | 43 | 24
Milligrams per decilitre*minute | -17414.0 (726.02) | 14236.9 (709.53) | 459.2 (947.50)
Statistical Analysis 1: Comparison: Semaglutide 1 mg vs Placebo; Test type: Other; p < 0.001, ANCOVA; Least Squares Mean Difference = -14696.1, 95% CI 2-sided [-17045.0 to -12347.3]
Statistical Analysis 2: Comparison: Tirzepatide 15 mg vs Placebo; Test type: Other; p < 0.001, ANCOVA; Least Squares Mean Difference = -17873.2, 95% CI 2-sided [-20239.0 to -15507.4]
Statistical Analysis 3: Comparison: Tirzepatide 15 mg vs Semaglutide 1 mg; Test type: Other; p = 0.002, ANCOVA; Least Squares Mean Difference = -3177.1, 95% CI 2-sided [-5194.3 to -1159.8]

4. Secondary Outcome: Change From Baseline in Hemoglobin A1c (HbA1c)
Description: HbA1c is the glycosylated fraction of hemoglobin A. HbA1c is measured primarily to identify average plasma glucose concentration over prolonged periods of time. LS mean was determined by mixed model repeated measures; (MMRM) model for post-baseline measures: Variable = Baseline + Treatment + Time + Treatment*Time (Type III sum of squares).
Time Frame: Baseline, Week 28
Population: All randomly assigned participants who received at least 1 dose of study drug and have evaluable data.
Measure: Least Squares Mean (Standard Error); unit: % of HbA1c
Arm/Group | Tirzepatide 15 mg | Semaglutide 1 mg | Placebo
Number analyzed (Participants) | 41 | 43 | 24
% of HbA1c | 2.05 (0.079) | -1.64 (0.078) | 0.29 (0.101)
Statistical Analysis 1: Comparison: Semaglutide 1 mg vs Placebo; Test type: Other; p < 0.001, Mixed Models Analysis; Least Squares Mean Difference = -1.93, 95% CI 2-sided [-2.18 to -1.67]
Statistical Analysis 2: Comparison: Tirzepatide 15 mg vs Placebo; Test type: Other; p < 0.001, Mixed Models Analysis; Least Squares Mean Difference = -2.33, 95% CI 2-sided [-2.58 to -2.08]
Statistical Analysis 3: Comparison: Tirzepatide 15 mg vs Semaglutide 1 mg; Test type: Other; p < 0.001, Mixed Models Analysis; Least Squares Mean Difference = -0.41, 95% CI 2-sided [-0.63 to -0.19]

5. Secondary Outcome: Change From Baseline in Total Insulin Secretion Rate During the 120-Minute Hyperglycemic Clamp (ISR0-120min)
Description: Total Insulin Secretion Rate During the 120-Minute Hyperglycemic Clamp (ISR0-120min) will be determined from C-peptide concentrations using the deconvolution technique. LS mean was determined by ANCOVA model for endpoint measures: log(Actual Measurement/Baseline) = log(Baseline) + Treatment (Type III sum of squares).
Time Frame: Baseline and Week 28
Population: All randomly assigned participants who received at least 1 dose of study drug and have evaluable data.
Measure: Least Squares Mean (Standard Error); unit: pmol/min/m^2
Arm/Group | Tirzepatide 15 mg | Semaglutide 1 mg | Placebo
Number analyzed (Participants) | 41 | 43 | 24
pmol/min/m^2 | 388.6 (20.17) | 286.6 (15.82) | 7.4 (7.15)
Statistical Analysis 1: Comparison: Semaglutide 1 mg vs Placebo; Test type: Other; p < 0.001, ANCOVA; Data were analysed with ANCOVA in log transformed data; Least Squares Mean Difference = 279.14, 95% CI 2-sided [245.10 to 313.18], Standard Error of Mean 17.366 — Data were analysed with ANCOVA in log transformed data. Results were converted back to original scale
Statistical Analysis 2: Comparison: Tirzepatide 15 mg vs Placebo; Test type: Other; p < 0.001, ANCOVA; Data were analysed with ANCOVA in log transformed data; Least Squares Mean Difference = 381.23, 95% CI 2-sided [339.29 to 423.17], Standard Error of Mean 21.399 — Data were analysed with ANCOVA in log transformed data. Results were converted back to original scale
Statistical Analysis 3: Comparison: Tirzepatide 15 mg vs Semaglutide 1 mg; Test type: Other; p < 0.001, ANCOVA; Data were analysed with ANCOVA in log transformed data; Least Squares Mean Difference = 102.09, 95% CI 2-sided [51.84 to 152.33], Standard Error of Mean 25.635 — Data were analysed with ANCOVA in log transformed data. Results were converted back to original scale

6. Secondary Outcome: Change From Baseline in Hyperinsulinemic Euglycemic Clamp M-value
Description: Hyperinsulinemic euglycemic clamp M-value is calculated from glucose infusion rate (GIR) over the last 30 minutes, corresponding to steady-state (+150 to +180 minutes), corrected for urine loss and space. LS mean was determined by ANCOVA model for endpoint measures: Variable = Baseline + Treatment (Type III sum of squares).
Time Frame: Baseline, Week 28
Population: All randomly assigned participants who received at least 1 dose of study drug and have evaluable data.
Measure: Least Squares Mean (Standard Error); unit: umol/min/kg [body weight]
Arm/Group | Tirzepatide 15 mg | Semaglutide 1 mg | Placebo
Number analyzed (Participants) | 41 | 39 | 24
umol/min/kg [body weight] | 19.2 (1.93) | 10.7 (1.99) | -0.6 (2.53)
Statistical Analysis 1: Comparison: Semaglutide 1 mg vs Placebo; Test type: Other; p < 0.001, ANCOVA; Least Squares Mean Difference = 11.3, 95% CI 2-sided [4.9 to 17.7]
Statistical Analysis 2: Comparison: Tirzepatide 15 mg vs Placebo; Test type: Other; p < 0.001, ANCOVA; Least Squares Mean Difference = 19.8, 95% CI 2-sided [13.4 to 26.1]
Statistical Analysis 3: Comparison: Tirzepatide 15 mg vs Semaglutide 1 mg; Test type: Other; p = 0.003, ANCOVA; Least Squares Mean Difference = 8.5, 95% CI 2-sided [3.0 to 14.0]

7. Secondary Outcome: Change From Baseline in Glucagon Concentration at Fasting
Description: Glucagon concentration was measured prior to sMMTT. LS mean was determined by ANCOVA model for endpoint measures: Variable = Baseline + Treatment (Type III sum of squares).
Time Frame: Baseline and Week 28
Population: All randomly assigned participants who received at least 1 dose of study drug and have evaluable data.
Measure: Least Squares Mean (Standard Error); unit: picomoles per litre (pmol/L)
Arm/Group | Tirzepatide 15 mg | Semaglutide 1 mg | Placebo
Number analyzed (Participants) | 40 | 40 | 22
picomoles per litre (pmol/L) | -3.6 (0.55) | -2.8 (0.55) | 0.8 (0.75)
Statistical Analysis 1: Comparison: Semaglutide 1 mg vs Placebo; Test type: Other; p < 0.001, ANCOVA; Least Squares Mean Difference = -3.6, 95% CI 2-sided [-5.5 to -1.8]
Statistical Analysis 2: Comparison: Tirzepatide 15 mg vs Placebo; Test type: Other; p < 0.001, ANCOVA; Least Squares Mean Difference = -4.5, 95% CI 2-sided [-6.3 to -2.6]
Statistical Analysis 3: Comparison: Tirzepatide 15 mg vs Semaglutide 1 mg; Test type: Other; p = 0.277, ANCOVA; Least Squares Mean Difference = -0.8, 95% CI 2-sided [-2.4 to 0.7]

8. Secondary Outcome: Change From Baseline in Glucagon Concentration at Postmeal
Description: Total AUC from time zero to 240 minutes after start of the meal [AUC0-240min]) during sMMTT. LS mean was determined by ANCOVA model for endpoint measures: Variable = Baseline + Treatment (Type III sum of squares).
Time Frame: Baseline and Week 28
Population: All randomly assigned participants who received at least 1 dose of study drug and have evaluable data.
Measure: Least Squares Mean (Standard Error); unit: (pmol/L)*min
Arm/Group | Tirzepatide 15 mg | Semaglutide 1 mg | Placebo
Number analyzed (Participants) | 40 | 39 | 22
(pmol/L)*min | -843.6 (86.26) | -502.0 (87.33) | -205.9 (116.31)
Statistical Analysis 1: Comparison: Semaglutide 1 mg vs Placebo; Test type: Other; p = 0.044, ANCOVA; Slope = -296.1, 95% CI 2-sided [-584.8 to -7.5]
Statistical Analysis 2: Comparison: Tirzepatide 15 mg vs Placebo; Test type: Other; p < 0.001, ANCOVA; Least Squares Mean Difference = -637.7, 95% CI 2-sided [-925.2 to -350.2]
Statistical Analysis 3: Comparison: Tirzepatide 15 mg vs Semaglutide 1 mg; Test type: Other; p = 0.006, ANCOVA; Least Squares Mean Difference = -341.6, 95% CI 2-sided [-585.2 to -97.9]

9. Secondary Outcome: Change From Baseline in Food Intake During Ad Libitum Meal
Description: Ad libitum meal served buffet-style. Food intake was recorded during a 45 minute period. The sum of the caloric breakdown (carbohydrates, protein, and fats) was calculated from the respective nutritional information of the food items. LS mean was determined by MMRM model for post-baseline measures: Variable = Baseline + Treatment + Time + Treatment*Time (Type III sum of squares).
Time Frame: Baseline, Week 28
Population: All randomly assigned participants who received at least 1 dose of study drug and have evaluable data.
Measure: Least Squares Mean (Standard Error); unit: kilocalorie (kcal)
Arm/Group | Tirzepatide 15 mg | Semaglutide 1 mg | Placebo
Number analyzed (Participants) | 41 | 43 | 24
kilocalorie (kcal) | -348.4 (34.59) | -284.1 (33.94) | -38.6 (45.17)
Statistical Analysis 1: Comparison: Semaglutide 1 mg vs Placebo; Test type: Other; p < 0.001, Mixed Models Analysis; Least Squares Mean Difference = -245.5, 95% CI 2-sided [-357.7 to -133.3]
Statistical Analysis 2: Comparison: Tirzepatide 15 mg vs Placebo; Test type: Other; p < 0.001, Mixed Models Analysis; Least Squares Mean Difference = -309.8, 95% CI 2-sided [-423.0 to -196.6]
Statistical Analysis 3: Comparison: Tirzepatide 15 mg vs Semaglutide 1 mg; Test type: Other; p = 0.187, Mixed Models Analysis; Least Squares Mean Difference = -64.3, 95% CI 2-sided [-160.3 to 31.7]

ADVERSE EVENTS:
Time Frame: Up to Week 32
Description: All randomly assigned participants who received at least 1 dose of study drug and have evaluable data.
Arm/Group | Placebo | Semaglutide 1 mg | Tirzepatide 15 mg
All-Cause Mortality (participants affected / at risk) | 0/28 | 0/44 | 0/45
Serious Adverse Events (participants affected / at risk) | 2/28 | 0/44 | 1/45
Other Adverse Events (participants affected / at risk) | 18/28 | 43/44 | 41/45
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=28) | Semaglutide 1 mg (N=44) | Tirzepatide 15 mg (N=45)
Acute myocardial infarction (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Subacute pancreatitis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Ureterolithiasis (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=28) | Semaglutide 1 mg (N=44) | Tirzepatide 15 mg (N=45)
Vertigo (Ear and labyrinth disorders) | 1 (1) | 1 (1) | 4 (4)
Abdominal distension (Gastrointestinal disorders) | 1 (1) | 5 (5) | 5 (5)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 2 (3) | 5 (5)
Abdominal pain upper (Gastrointestinal disorders) | 3 (3) | 4 (6) | 5 (5)
Constipation (Gastrointestinal disorders) | 0 (0) | 8 (10) | 6 (6)
Diarrhoea (Gastrointestinal disorders) | 6 (8) | 13 (17) | 9 (10)
Dyspepsia (Gastrointestinal disorders) | 2 (3) | 14 (23) | 3 (3)
Eructation (Gastrointestinal disorders) | 0 (0) | 8 (8) | 8 (9)
Nausea (Gastrointestinal disorders) | 7 (8) | 13 (22) | 11 (22)
Vomiting (Gastrointestinal disorders) | 1 (1) | 5 (10) | 3 (3)
Asthenia (General disorders) | 0 (0) | 3 (3) | 3 (3)
Early satiety (General disorders) | 6 (6) | 12 (12) | 16 (16)
Fatigue (General disorders) | 2 (2) | 10 (11) | 5 (6)
Injection site haematoma (General disorders) | 12 (20) | 12 (21) | 12 (21)
Injection site pain (General disorders) | 2 (4) | 3 (3) | 1 (1)
Nasopharyngitis (Infections and infestations) | 3 (3) | 8 (14) | 7 (8)
Lipase increased (Investigations) | 2 (2) | 2 (2) | 5 (7)
Abnormal loss of weight (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 3 (3)
Decreased appetite (Metabolism and nutrition disorders) | 7 (7) | 31 (34) | 27 (29)
Back pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 2 (2) | 3 (3)
Dizziness (Nervous system disorders) | 0 (0) | 2 (2) | 3 (4)
Headache (Nervous system disorders) | 5 (5) | 7 (11) | 4 (5)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2020-06-10): https://cdn.clinicaltrials.gov/large-docs/53/NCT03951753/Prot_000.pdf
  • Statistical Analysis Plan (2021-05-27): https://cdn.clinicaltrials.gov/large-docs/53/NCT03951753/SAP_001.pdf